CLINICAL TRIAL: NCT04487535
Title: The Relationship Between Preoperative Serum Cytokine Level and Lenght of Stay in Hospital, Postoperative Pain Intensity, Functional Status, Joint Position Sense and X Ray Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Kübra Canli, Karadeniz Technical University, Karadeniz Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Karadeniz Technique Unıversty
Record Dates: First submitted 2020-07-16; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2018-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Cytokines; Proprioception; Pain; Functional Status; Lenght of Stay in hospital
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Total Knee Arthroplasty Surgery (Other): Surgery performed by one orthopedic surgeon
  Interventions: Other: Cytokine level

INTERVENTIONS:
Other: Cytokine level — Serum cytokine level will be measured before surgery, 72nd after surgery and 6 weeks after surgery

SUMMARY:
Serum cytokines was assosiated with symptoms and progression of osteoartritis. It is unknown whether these cytokines have a predictive role on severity of symptoms after total knee arthroplasty (TKA) or not. The aim of this study is to investigate the relationships between the preoperative serum cytokine level (SCL) and lenght of stay in hospital, postoperative pain intensity, functional status, joint position sense and X ray.

Grade 4 osteoartritis degeneration who intern the hospital for total knee arthroplasty surgery. Serum Cytokine Levels (IL-6, TNFα, IL-1β) will be assessed before surgery. Pain intensity at rest/activity and valgite angle will be evaluated before surgery, postoperative 72 hour and postoperative 6 weeks. Functional status and joint position sense will be assessed before surgery and 6 weeks after surgery. Lenght of stay in hospital (LOS) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 45-75
2. were scheduled for unilateral or bilateral TKA
3. were diagnosed of OA with a severity Grade 4 according to the Kellgren-Lawrence (KL) classification.

Exclusion Criteria:

1. neuropathic pain
2. presurgery for same lower extremity
3. vascular disease
4. any chronic disease related to kidney, heart, liver
5. cancer
6. chronic inflammatory disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pain intensty | pain intensity will be evaluated. It will determined pain intensity alteration from 2 weeks before surgery and at 72 hours and at 6 weeks following surgery
  Rest and activity pain intensity will be evaluated by using 100 mm vertical line Visual Anolog Scale (VAS). Zero meet no pain, 10 unbearable pain

SECONDARY OUTCOMES:
Functional Status | Functional status will be assessed before surgery and 6 weeks after surgery
  Turkish version of Western Ontario McMaster University Osteoarthritis Index (WOMAC) scale will be used to evaluate functional status. The WOMAC is a self reported funtional assessment scale consisting of 24 items which responded on Likert type scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme), with higher score indicating more difficulty
Joint Position Sense | It will be evaluated before surgery and 6 weeks after surgery
  Joint positon sense will be evaluated by using a digital goniometer. Each patient will be asked to sat in a erect pack position on the chair with knee relaxed in 90 º flexion noticing that popliteal fossa was not in contact with end edge of the chair. A digital goniometer will be placed at the lateral aspect of the knee, with moveable arm in the course of midline of the lateral malleolus and stationary arm along the midline of the femur. The knee will be moved passively by examiner slowly from initial position (90º flexion) to final predetermined three angle (35º, 55º, 70º), hold final positon for 5 second and then return to initial position with same speed. After instruction the procedure, patients will be ask to extend the knee actively for each angle. This procedure will be repeated three times for each angle.
X-Ray | X-ray evaluated before surgery, 72 hour after surgery and 6 weeks ater surgery
  To measure valgus angle, standart anteroposterior (AP) X ray view was obtained from patients in standing position and without shoes. The angle between femoral axis which indicate a line drawn from femoral head to femoral intercondylar notch and tibial axis which describe a line from the center of the talus bone to the center of the tibial spine was measured by orthopedics
Serum Cytokine Level | Venous blood sample was collected 2 weeks before surgery
  Five-milliliter blood samples from each individual were placed into vacutainer tubes without anticoagulant. These were then centrifuged at 1800 g for 10 minutes. Serum samples were stored at -80°C until being used for measurements. Serum IL- 6, TNF-α ve IL-1β levels were determined using commercial sandwich-ELISA kits. The absorbance of the samples was measured at a 450 nm wavelength on a VERSA (designed by Molecular Devices in California, USA) micro plate reader. The results were expressed as pg/ mL. The coefficients of variation (CV) of this ELISA method were6.69% for IL-6, 6.62% for TNF alfa and 6.72% for IL-1beta.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Universty, Ankara, Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No